## DynaSSaur:

## **Consent form: Control Group**

| Full study name: | | Dynamic Chest X-ray with Simultaneous Spirometry | |
|---|---|---|---|
| IRAS: | | 322890 | |
| Principal investigator:<br>Co-investigators: | | Dr David Green<br>Professor Martin Walshaw<br>Dr Dilip Nazareth<br>Dr Freddy Frost | |
| | | | Please<br>initial box |
| 1. | <ol> <li>I confirm that I have read the Participant Information Sheet dated 20/09/2023 (version 3.1) for the above study. I have had the opportunity to consider the information, ask questions, and have had these answered satisfactorily.</li> </ol> | | |
| 2. | I understand that my participation is voluntary and that I am free to withdraw at any time without giving any reason, and without my medical care or legal rights being affected. | | |
| 3. | I understand that my data will be stored securely on NHS servers or within locked areas of LHCH, in line with NHS data protection regulations, GDPR (General Data protection regulation) and DPA (Data Protection Act 2018). GDPR and The DPA are designed to regulate how data should be handled appropriately to protect personalised information. | | |
| 4. | | draw from this study, the researchers may keep my information for nely keep this information for up to 20 years. | |

Version 3.1 Date 20/09/2023

| <ol> <li>I understand that the information and data collected during the study may be looked at by members of the study team where it is relevant to me taking part in this research. I give permission for these individuals to have access to this data collected.</li> <li>I understand that the information collected about me will be used to support other research in the future and may be shared anonymously with other researchers.</li> <li>I understand that the information held and maintained by LHCH may be used to help contact me or provide information about my health status. I understand that as part of this process, my GP may be contacted if there is clinical information that they need to know or act upon.</li> <li>I agree to take part in the above study, which will involve an interview to establish background medical history. It will also involve me attending LHCH for a dynamic chest X-ray and spirometry (breathing tests).</li> <li>I understand that any information I write in the questionnaire 'free text' box may be published, in a completely anonymous form, by the study team.</li> </ol> | Name of participant | | Date | Signature |
|---|---|---|---|---|
| <ul> <li>members of the study team where it is relevant to me taking part in this research. I give permission for these individuals to have access to this data collected.</li> <li>6. I understand that the information collected about me will be used to support other research in the future and may be shared anonymously with other researchers.</li> <li>7. I understand that the information held and maintained by LHCH may be used to help contact me or provide information about my health status. I understand that as part of this process, my GP may be contacted if there is clinical information that they need to know or act upon.</li> <li>8. I agree to take part in the above study, which will involve an interview to establish background medical history. It will also involve me attending LHCH for a dynamic chest X-ray and spirometry (breathing tests).</li> <li>9. I understand that any information I write in the questionnaire 'free text' box may be published,</li> </ul> | | and completely unonymou | | |
| <ul> <li>members of the study team where it is relevant to me taking part in this research. I give permission for these individuals to have access to this data collected.</li> <li>6. I understand that the information collected about me will be used to support other research in the future and may be shared anonymously with other researchers.</li> <li>7. I understand that the information held and maintained by LHCH may be used to help contact me or provide information about my health status. I understand that as part of this process, my GP may be contacted if there is clinical information that they need to know or act upon.</li> <li>8. I agree to take part in the above study, which will involve an interview to establish background medical history. It will also involve me attending LHCH for a dynamic chest X-ray</li> </ul> | 9. | | | |
| <ul> <li>members of the study team where it is relevant to me taking part in this research. I give permission for these individuals to have access to this data collected.</li> <li>6. I understand that the information collected about me will be used to support other research in the future and may be shared anonymously with other researchers.</li> <li>7. I understand that the information held and maintained by LHCH may be used to help contact me or provide information about my health status. I understand that as part of this process,</li> </ul> | 8. | background medical history. It will also involve me attending LHCH for a dynamic chest X-ray | | |
| members of the study team where it is relevant to me taking part in this research. I give permission for these individuals to have access to this data collected. 6. I understand that the information collected about me will be used to support other research in | 7. | me or provide information about my health status. I understand that as part of this process, | | |
| members of the study team where it is relevant to me taking part in this research. I give | 6. | | | |
| | U. | | | |

One copy of this consent form is to be stored securely in the Site Investigator File.

One copy of this consent form is to be provided to the participant.

Version 3.1 Date 20/09/2023